CLINICAL TRIAL: NCT04437797
Title: Soft Tissue Outcomes of Badly Broken-down Teeth Treated With Surgical Extrusion Compared With Immediate Implant Placement: A Randomized Controlled Trial
Brief Title: Soft Tissue Outcomes of Badly Broken-down Teeth Treated With Surgical Extrusion Compared With Immediate Implant Placement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ismail Tarek Mansour, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21/4/2020
Record Dates: First submitted 2020-06-15; First posted 2020-06-18 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Broken Teeth
MeSH Terms: conditions — Tooth Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical Extrusion (Experimental): The next step will be atraumatic extraction which will be initiated by using straight periotome until it is sufficiently luxated and gently pulled out to the amount of sufficient ferrule effect without encroaching the biological width. 90- or 180-degrees rotation of the tooth will be done if needed. The tooth will be supported from palatal side, etching will be done using 37% phosphoric acid, rinsing, drying, bonding agent and then application of 3M Filtek flowable composite on rounded 16mm stainless steel wire for splinting in the middle of the tooth without extension of flowable composite neither to the mesial nor to the distal. This procedure should be followed by occlusal adjustment if needed. Splint will be removed after 2 weeks.
  Interventions: Procedure: Surgical Extrusion
- Immediate Implant Placement (Active Comparator): The patient is anaesthetized. Atraumatic extraction of the badly broken-down teeth will be performed using peroiotome. Luxation should be done mesiodistally and not buccolingually, 11 to avoid damaging the buccal plate. After tooth removal, a curette is used to confirm that the location of the buccal plate is intact. Standard drilling procedures are performed according to the manufacturer's instructions. Then the implant is placed in the prepared site. Temporization should be done using composite 3M Filtek Z250 XT material. Finally, a porcelain fused to zirconia crown will be performed. Jumping gap occurring subsequent to atraumatic extraction and immediate implant placement more than 2 mm will be grafted using Xenograft.
  Interventions: Procedure: Immediate Implant Placement

INTERVENTIONS:
Procedure: Surgical Extrusion — The next step will be atraumatic extraction which will be initiated by using straight periotome until it is sufficiently luxated and gently pulled out to the amount of sufficient ferrule effect without encroaching the biological width. 90- or 180-degrees rotation of the tooth will be done if needed. The tooth will be supported from palatal side, etching will be done using 37% phosphoric acid, rinsing, drying, bonding agent and then application of 3M Filtek flowable composite on rounded 16mm stainless steel wire for splinting in the middle of the tooth without extension of flowable composite neither to the mesial nor to the distal. This procedure should be followed by occlusal adjustment if needed. Splint will be removed after 2 weeks.
  Arms: Surgical Extrusion
Procedure: Immediate Implant Placement — The patient is anaesthetized. Atraumatic extraction of the badly broken-down teeth will be performed using peroiotome. Luxation should be done mesiodistally and not buccolingually, 11 to avoid damaging the buccal plate. After tooth removal, a curette is used to confirm that the location of the buccal plate is intact. Standard drilling procedures are performed according to the manufacturer's instructions. Then the implant is placed in the prepared site. Temporization should be done using composite 3M Filtek Z250 XT material. Finally, a porcelain fused to zirconia crown will be performed. Jumping gap occurring subsequent to atraumatic extraction and immediate implant placement more than 2 mm will be grafted using Xenograft.
  Arms: Immediate Implant Placement

SUMMARY:
Many patients suffer from badly decayed anterior teeth mostly in young age, causing esthetics and functional issues. This may be due to more than cause as fights, contact sports, accidents and falls.

However; implant placement might not be the treatment of choice in some situations such as: medically compromised patients with absolute contraindications for implant placement or requiring extensive augmentation procedures, growing patients, patients with financial limitations, in addition to patients living in rural areas with no access for CBCT machines.

Moreover, clinicians must be aware of cost-to-benefit ratios when attempting to recommend a specific treatment modality, especially in patients having financial limitations.

Regarding the aforementioned conditions, surgical extrusion might be considered a cost-effective 'often overlooked' alternative compared to immediate single-tooth implant placement. Regarding healing time, cost, soft and hard tissue outcomes, surgical extrusion may be a good alternative yielding better soft tissue results as we preserve the natural tooth with the whole periodontium.

ELIGIBILITY:
Inclusion Criteria:

1. Patients at 20-40 years old and have no history of periodontal disease. (periodontally healthy patients)
2. Single rooted teeth; should be single with adjacent intact or restored neighboring teeth. More than one tooth may be included in the same arch.
3. More than 1:1 crown root ratio, so that the crown to root ratio is 1:1 after extrusion and restoration

Exclusion Criteria:

1. Badly broken-down teeth with active signs of infection.
2. Teeth with vertical root fracture.
3. Teeth with severely tapered root.
4. Diabetic patients, assessed by measuring glycosylated hemoglobin (HbA1c). Patients with an HbA1c level greater than 8 will be excluded.
5. Potentially uncooperative patients who are not willing to go through the proposed interventions.
6. Moderate-to-heavy daily smokers* (who report consuming at least 11 cigarettes/day). 9
7. History of radiation therapy and/or chemotherapy to the head and neck, or bone augmentation to implant site.
8. Labial cortical bone fenestration diagnosed from CBCT.
9. Patients with systemic disease that may affect normal healing.
10. Psychiatric problems, emotional instability, and unrealistic esthetic demands.
11. Bruxism.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Soft tissue outcome | 12 months
  Pink esthetic score: 0-1-2 scoring system, 0 being the lowest, 2 being the highest value

SECONDARY OUTCOMES:
Survival | 12 months
  Tooth and Implant survival (binary)

CONTACTS AND LOCATIONS:
Overall Officials: Ismail T Mansour, B.D.S., Principal Investigator — Cairo University

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Bastone EB, Freer TJ, McNamara JR. Epidemiology of dental trauma: a review of the literature. Aust Dent J. 2000 Mar;45(1):2-9. doi: 10.1111/j.1834-7819.2000.tb00234.x. PMID 10846265
- [Background] Gomez-de Diego R, Mang-de la Rosa Mdel R, Romero-Perez MJ, Cutando-Soriano A, Lopez-Valverde-Centeno A. Indications and contraindications of dental implants in medically compromised patients: update. Med Oral Patol Oral Cir Bucal. 2014 Sep 1;19(5):e483-9. doi: 10.4317/medoral.19565. PMID 24608222
- [Background] Clokie CM, Yau DM, Chano L. Autogenous tooth transplantation: an alternative to dental implant placement? J Can Dent Assoc. 2001 Feb;67(2):92-6. PMID 11253297
- [Background] Mamoun JS. On the ferrule effect and the biomechanical stability of teeth restored with cores, posts, and crowns. Eur J Dent. 2014 Apr;8(2):281-286. doi: 10.4103/1305-7456.130639. PMID 24966784
- [Background] Walsh JS, Kafrawy A, Roche JR. The effect of apical modification on the vitality of replanted permanent monkey teeth. ASDC J Dent Child. 1978 Mar-Apr;45(2):146-50. No abstract available. PMID 96161
- [Background] Nugala B, Kumar BS, Sahitya S, Krishna PM. Biologic width and its importance in periodontal and restorative dentistry. J Conserv Dent. 2012 Jan;15(1):12-7. doi: 10.4103/0972-0707.92599. PMID 22368328
- [Background] Bach N, Baylard JF, Voyer R. Orthodontic extrusion: periodontal considerations and applications. J Can Dent Assoc. 2004 Dec;70(11):775-80. PMID 15588553
- [Background] Singh M, Kumar L, Anwar M, Chand P. Immediate dental implant placement with immediate loading following extraction of natural teeth. Natl J Maxillofac Surg. 2015 Jul-Dec;6(2):252-5. doi: 10.4103/0975-5950.183864. PMID 27390509
- [Background] Belser UC, Grutter L, Vailati F, Bornstein MM, Weber HP, Buser D. Outcome evaluation of early placed maxillary anterior single-tooth implants using objective esthetic criteria: a cross-sectional, retrospective study in 45 patients with a 2- to 4-year follow-up using pink and white esthetic scores. J Periodontol. 2009 Jan;80(1):140-51. doi: 10.1902/jop.2009.080435. PMID 19228100
- [Background] Papaspyridakos P, Chen CJ, Singh M, Weber HP, Gallucci GO. Success criteria in implant dentistry: a systematic review. J Dent Res. 2012 Mar;91(3):242-8. doi: 10.1177/0022034511431252. Epub 2011 Dec 8. PMID 22157097
- [Background] Misch CE, Perel ML, Wang HL, Sammartino G, Galindo-Moreno P, Trisi P, Steigmann M, Rebaudi A, Palti A, Pikos MA, Schwartz-Arad D, Choukroun J, Gutierrez-Perez JL, Marenzi G, Valavanis DK. Implant success, survival, and failure: the International Congress of Oral Implantologists (ICOI) Pisa Consensus Conference. Implant Dent. 2008 Mar;17(1):5-15. doi: 10.1097/ID.0b013e3181676059. PMID 18332753
- [Background] Annibali S, Bignozzi I, La Monaca G, Cristalli MP. Usefulness of the aesthetic result as a success criterion for implant therapy: a review. Clin Implant Dent Relat Res. 2012 Mar;14(1):3-40. doi: 10.1111/j.1708-8208.2009.00234.x. Epub 2009 Aug 6. PMID 19673953
- [Background] Sheng L, Silvestrin T, Zhan J, Wu L, Zhao Q, Cao Z, Lou Z, Ma Q. Replacement of severely traumatized teeth with immediate implants and immediate loading: literature review and case reports. Dent Traumatol. 2015 Dec;31(6):493-503. doi: 10.1111/edt.12201. Epub 2015 Jul 14. PMID 26176171